CLINICAL TRIAL: NCT06459804
Title: Effects of Electro Dry Needling Versus Dry Needling on Pain, Muscle Strength, and Range of Motion in Patients With Levator Scapulae Syndrome
Brief Title: Effects of Electro Dry Needling Versus Dry Needling in Levator Scapulae Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCRS/1021 Aqsa
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Neck Syndrome
Keywords: neck pain; disability; muscle strength; Range of Motion
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Electro Dry Needling (Experimental): Group A: will receive Electro Dry Needling along with conventional physiotherapy. The parameters for Electro dry needling will be needles of 30×0.25 mm, 50×0.25 mm sizes, Frequency 80-100 Hz, Duration 10-20 minutes and intensity as tolerated.
  Interventions: Procedure: Electro Dry Needling
- Group B: Dry Needling (Active Comparator): Group B will receive Dry Needling along with conventional Physiotherapy in which parameters will be dry needles will be 30×0.25 and 50×0.25 mm sizes, Frequency 80-100 Hz, Duration 10-20 minutes and intensity as tolerated.
  Interventions: Procedure: Dry Needling

INTERVENTIONS:
Procedure: Electro Dry Needling — Standard Physiotherapy:
  It will include Hot pack (10 min), Stretching of levator scapulae (3 times with 30 seconds hold), Scapular stabilization exercises (10 times with 5 seconds hold).
  Scapular Stabilization exercises will be comprised of four exercise programs. The participants will sit on the knees in 90° flexion position, and a Swiss ball will be propped up between the stomach and chest.
  Arms: Group A: Electro Dry Needling
Procedure: Dry Needling — Dry Needling
  Arms: Group B: Dry Needling

SUMMARY:
Mechanical neck pain is posteriorly occurring non-specific pain that originates from the superior nuchal line and extends to the first thoracic vertebrae. It is exacerbated by sustained neck postures, neck movements or cervical muscle palpation. The aim of study will be to compare the effects of Electro Dry Needling and Dry Needling on pain, muscle strength, disability and range of motion in patients with Levator Scapulae Syndrome.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Shalamar Hospital, (SIHS Physiotherapy Clinic Lahore) through convenience sampling technique on 30 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will receive Electro Dry Needling along with conventional physiotherapy in which parameters for Electro dry needling will be needles of 30×0.25 mm, 50×0.25 mm sizes, Frequency 80-100 Hz, Duration 10-20 minutes and intensity as tolerated and Group B will receive Dry Needling along with conventional Physiotherapy in which parameters will be dry needles will be 30×0.25 and 50×0.25 mm sizes. Standard Physiotherapy will include a Hot pack (10 min), Stretching of levator scapulae (3 times with 30 second hold), and Scapular stabilization exercises (10 times with 5 second hold).There will be 3 sessions per week, Needling in both groups will be for performed 2 times per week for total 3rd week of treatment comprising of 6 sessions, 3rd session will comprise of standard physical therapy. Pre and Post treatment measures will be recorded.Outcome measures will be conducted through pain, *muscle strength,* disability and range of motion questionnaire. Data will be analyzed during *SPSS software version 25.After assessing the normality of data by the Shapiro-Wilk test, it will be decided whether a parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges of 18-45 years
* Both genders, males and females
* Positive Levator Scapular length Test (7)
* Positive Simon's criteria for Levator scapulae
* Neck pain -NPRS < 7 (8)
* Neck and upper back pain for at least 3months.
* Examination - Increased muscle tone and tenderness at neck and upper back
* Reduced ROM-Side flexion and Rotation of neck
* Non traumatic unilateral mechanical neck pain of three or more months of duration, presenting an latent MTrP in the levator scapulae muscle on the painful side

Exclusion Criteria:

* Neuropathies
* Radiated pain towards the arm
* Vertebral fractures
* Traumatic neck injury
* whiplash injury (9)
* previous surgical procedures in the cervical spine
* Previous cognitive and functional disorders
* psychological disorders (mood and psychotic disorders such as schizophrenia, depression,and anxiety disorders),
* Fibromyalgia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Numeric pain rate scale (NPRS) | upto 3 weeks
  The NPRS is a segmented numeric version in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. the NPRS is anchored by terms describing pain severity extremes.
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Neck Disability index (NDI) | upto 3 weeks
  The results of this questionnaire have been utilized to evaluate the disability. It consists of 10 items: 7 linked to activities of daily living, 2 to pain, and 1 to concentration. From 0 to 5, each item received a score. Higher scores corresponded to more disability, and the total score was reported as a percentage.
Universal Goniometer | upto 3 weeks
  An instrument called a goniometer is used to measure a joint's range of motion. Physical therapists typically use a goniometer to measure a range of motion. At the initial evaluation, the therapist can determine the possible range of motion using a goniometer .
  Range of motion: Side flexion and Rotation of neck measured with Goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Aqsa Wahid, MSPT*, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Aqsa Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-de-Miguel S, Pecos-Martin D, Larroca-Sanz T, Sanz-de-Vicente B, Garcia-Montes L, Fernandez-Matias R, Gallego-Izquierdo T. Short-Term Effects of PENS versus Dry Needling in Subjects with Unilateral Mechanical Neck Pain and Active Myofascial Trigger Points in Levator Scapulae Muscle: A Randomized Controlled Trial. J Clin Med. 2020 Jun 1;9(6):1665. doi: 10.3390/jcm9061665. PMID 32492884
- [Background] Hernandez-Secorun M, Abenia-Benedi H, Borrella-Andres S, Marques-Garcia I, Lucha-Lopez MO, Herrero P, Iguacel I, Tricas-Moreno JM, Hidalgo-Garcia C. Effectiveness of Dry Needling in Improving Pain and Function in Comparison with Other Techniques in Patients with Chronic Neck Pain: A Systematic Review and Meta-Analysis. Pain Res Manag. 2023 Aug 23;2023:1523834. doi: 10.1155/2023/1523834. eCollection 2023. PMID 37664417
- [Background] ALchlaihawi A, Tajali SB, Malmir K, Mahdi TS (2023) Effects of Dry Needling and Dry Needling Combined with Electrical Stimulation on Pain and Function in Patients with Subacute Musculoskeletal Neck Pain Following Myofascial Trigger Points. History of Medicine 9(1): 1845-1858. https://doi.org/10.17720/24095834.v9.1.2023.237
- [Background] Song Young-mun, Weon Jong-hyuck, Jung Do-young. Reliability of a New Test of Levator Scapula Muscle Length. J Musculoskelet Sci Technol 2019;3(1):1-6. https://doi.org/10.29273/jmst.2019.3.1.1
- [Background] Gattie E, Cleland JA, Snodgrass S. The Effectiveness of Trigger Point Dry Needling for Musculoskeletal Conditions by Physical Therapists: A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2017 Mar;47(3):133-149. doi: 10.2519/jospt.2017.7096. Epub 2017 Feb 3. PMID 28158962
- [Background] Liu L, Huang QM, Liu QG, Ye G, Bo CZ, Chen MJ, Li P. Effectiveness of dry needling for myofascial trigger points associated with neck and shoulder pain: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):944-55. doi: 10.1016/j.apmr.2014.12.015. Epub 2015 Jan 7. PMID 25576642